CLINICAL TRIAL: NCT00176852
Title: Allogeneic Hematopoietic Stem Cell Transplant for Patients With High Risk Hemoglobinopathy Using a Preparative Regimen to Achieve Stable Mixed Chimerism
Brief Title: Stem Cell Transplant for Hemoglobinopathy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT2002-07; 0206M26241 (Other: IRB, University of Minnesota); NCT00005897 (obsolete NCT alias)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2017-05-09 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Sickle Cell Disease; Thalassemia; Severe Congenital Neutropenia; Diamond-Blackfan Anemia; Shwachman-Diamond Syndrome
Keywords: high risk hemoglobinopathy; stem cell transplant; donor lymphocyte infusion; transfusion dependent; stem cell donor; cord blood; marrow; transfusion dependent non-malignant hematologic disorders
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia; Neutropenia, Severe Congenital, Autosomal Recessive 3; Anemia, Diamond-Blackfan; Shwachman-Diamond Syndrome | interventions — Busulfan; fludarabine; fludarabine phosphate; Cyclophosphamide; Antilymphocyte Serum; Granulocyte Colony-Stimulating Factor; Alemtuzumab; Whole-Body Irradiation; Bone Marrow Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RIC Bu/Flu (A) (discontinued) (Other): Full Preparative Regimen for subjects with matched donors using Busulfan on Day -8 and -7, Fludarabine on Day -6 through -2, antithymocyte globulin (ATG) on Day -2 through -1, total lymphoid radiation (TLI) on Day -1, stem cell infusion on Day 0.
  Interventions: Drug: Busulfan, Fludarabine, ATG, TLI
- MA Bu/Cy (B) (Experimental): Myeloablative Preparative Regimen for subjects with HLA identical sibling donors consists of Busulfan on day -9 through -6, Cyclophosphamide on day -5 through -2, ATG on day -3 through -1, stem cell infusion on Day 0 and Granulocyte Colony Stimulating Factor on day -3 until ANC >2500 x 2 days.
  Interventions: Drug: Busulfan, Cyclophosphamide, ATG, GCSF; Radiation: Total Body Irradiation; Procedure: Stem cell infusion
- RIC Cy/Flu/TBI (A2) (Experimental): Patients with sickle cell disease or thalassemia who do not have an HLA-identical sibling donor or who has pre-existing organ dysfunction making myeloablative condition ineligible will receive Campath on day -10 through -6, Cyclophosphamide on day -7, Fludarabine on day -6 through -2, total body irradiation (TBI) on day -1, stem cell infusion on Day 0.
  Interventions: Drug: Campath, Fludarabine, Cyclophosphamide; Radiation: Total Body Irradiation; Procedure: Stem cell infusion

INTERVENTIONS:
Drug: Busulfan, Fludarabine, ATG, TLI — Busulfan 0.8 mg/kg/dose intravenous (IV) Days -8 and -7 Fludarabine 35 mg/m2 IV Days -6 through -2 Antithymocyte globulin (ATG) 30 mg/kg IV Days -2 and -1 Total lymphoid radiation 300 cGy
  Other Names: Busulfex; Fludara; ATG; Total lymphoid Irradiation
  Arms: RIC Bu/Flu (A) (discontinued)
Drug: Busulfan, Cyclophosphamide, ATG, GCSF — Busulfan 0.8 mg/kg/dose intravenous (IV) Days -9 through -6 Cyclophosphamide 50 mg/kg IV Days -5 through -2 ATG 30 mg/kg IV Day -1 GCSF 5 mcg/kg/day IV until ANC >2500 x 2 days.
  Other Names: Busulfex; Cytoxan; antithymocyte globulin; granulocyte colony-stimulating factor
  Arms: MA Bu/Cy (B)
Drug: Campath, Fludarabine, Cyclophosphamide — Receives Campath-1H 0.2 mg/kg Days -10 through -6, Fludarabine 35 mg/m2 intravenous (IV) Days -6 through -2, total body irradiation (TBI) 300 cGy Day -1.
  Other Names: Fludara; alemtuzumab; Cytoxan
  Arms: RIC Cy/Flu/TBI (A2)
Radiation: Total Body Irradiation — 300 cGY Day -1
  Other Names: TBI
  Arms: MA Bu/Cy (B); RIC Cy/Flu/TBI (A2)
Procedure: Stem cell infusion — Given Day 0
  Other Names: bone marrow transplant
  Arms: MA Bu/Cy (B); RIC Cy/Flu/TBI (A2)

SUMMARY:
This study tests the clinical outcomes of one of two preparative regimens (determined by available donor source) in patients with non-malignant hemoglobinopathies. The researchers hypothesize that these regimens will have a positive effect on post transplant engraftment and the incidence of graft-versus-host-disease.

Regimen A2 has replaced Regimen A in this study. Two patients were treated on Regimen A but did not have evidence of initial engraftment thus triggering the stopping rule for that arm of this study.

DETAILED DESCRIPTION:
Prior to transplantation, subjects will receive either:

Cyclophosphamide, Fludarabine, Campath, Total body irradiation (TBI)

Or

Busulfan, Cyclophosphamide, antithymocyte globulin (ATG), granulocyte colony-stimulating factor (GSCF)

These drugs (and the radiation) are being given to help the new stem cells take and grow. On the day of transplantation, subjects will receive stem cells transfused via intravenous (IV) catheter.

After stem cell transplantation, subjects will be given cyclosporine-A and mycophenolate (MMF)/or Methylprednisone/or Methotrexate to reduce the risk of graft-versus-host disease, the complication that occurs when the donor's stem cells react against the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Sickle Cell Disease/Thalassemia (SCD/THAL) 0-50 years of age with an acceptable stem cell donor and disease characteristic defined by the following:

  * Stroke, central nervous system (CNS) hemorrhage or a neurologic event lasting longer than 24 hours, or abnormal cerebral magnetic resonance imaging (MRI) or cerebral arteriogram or MRI angiographic study and impaired neuropsychological testing
  * Acute chest syndrome with a history of recurrent hospitalizations or exchange transfusions
  * Recurrent vaso-occlusive pain 3 or more episodes per year for 3 years or more years or recurrent priapism,
  * Impaired neuropsychological function and abnormal cerebral MRI scan
  * Stage I or II sickle lung disease,
  * Sickle nephropathy (moderate or severe proteinuria or a glomerular filtration rate [GFR] 30-50% of the predicted normal value)
  * Bilateral proliferative retinopathy and major visual impairment in at least one eye
  * Osteonecrosis of multiple joints with documented destructive changes
  * Requirement for chronic transfusions but with red blood cell (RBC) alloimmunization >2 antibodies during long term transfusion therapy
* Patients with transfusion dependent alpha- or beta-thalassemia 0-35 years of age with an acceptable stem cell donor as defined in the criteria in section above.
* Patients with other non-malignant hematologic disorders that are transfusion-dependent or involve other potentially life-threatening cytopenias (including but not limited to Severe Congenital Neutropenia, Diamond-Blackfan Anemia and Shwachman-Diamond Syndrome) who are 0-35 years of age with an acceptable stem cell donor
* Second Transplants

  * Patients with sickle cell disease or thalassemia who have failed to engraft or have autologous recovery after a myeloablative SCT regimen or non-myeloablative regimen are eligible for this protocol.
  * Regimen A2 will be utilized for patients with sickle cell disease or thalassemia who do not have an HLA-identical sibling donor or for any patient who has pre-existing organ dysfunction making them ineligible for a myeloablative preparative regimen.
  * Regimen B will be utilized for patients with sickle cell disease or thalassemia who have an HLA-identical sibling donor.
  * Patients must meet above criteria.
  * If the patient has received prior radiation therapy, eligibility to receive additional radiation therapy must be determined by Dr. Dusenbery
  * If first transplant was a non-myeloablative regimen, the second transplant can occur at any time
  * If the first transplant was a myeloablative regimen, then the second transplant must be > 6 months from the first transplant

Exclusion Criteria:

* Patients with one or more of the following:
* Karnofsky or Lansky performance score <70
* Acute hepatitis or evidence of moderate or severe portal fibrosis or cirrhosis on biopsy
* Stage III-IV lung disease
* GFR<30% predicted
* Pregnant or lactating females
* Active serious infection whereby patient has been on intravenous antibiotics for one week prior to study entry. Any patient with AIDS or ARC or HIV seropositivity
* Psychologically incapable of undergoing bone marrow transplant (BMT) with associated strict isolation or documented history of medical non-compliance
* Patients not able to receive total lymphocytic irradiation (TLI) due to prior radiation therapy

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2002-06; Primary Completion 2014-03 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Angela Smith, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Conditioning (Discontinued / A): Full Preparative Regimen for subjects with matched donors using Busulfan on Day -8 and -7, Fludarabine on Day -6 through -2, antithymocyte globulin (ATG) on Day -2 through -1, total lymphoid radiation (TLI) on Day -1, stem cell infusion on Day 0.
  Busulfan, Fludarabine, ATG, TLI: Busulfan 0.8 mg/kg/dose intravenous (IV) Days -8 and -7 Fludarabine 35 mg/m2 IV Days -6 through -2 Antithymocyte globulin (ATG) 30 mg/kg IV Days -2 and -1 Total lymphoid radiation 300 cGy
- Busulfan Conditioning (B): Myeloablative Preparative Regimen for subjects with HLA identical sibling donors consists of Busulfan on day -9 through -6, Cyclophosphamide on day -5 through -2, ATG on day -3 through -1, stem cell infusion on Day 0 and Granulocyte Colony Stimulating Factor on day -3 until ANC >2500 x 2 days.
  Busulfan, Cyclophosphamide, ATG, GCSF: Busulfan 0.8 mg/kg/dose intravenous (IV) Days -9 through -6 Cyclophosphamide 50 mg/kg IV Days -5 through -2 ATG 30 mg/kg IV Day -1 GCSF 5 mcg/kg/day IV until ANC >2500 x 2 days.
  Total Body Irradiation: 300 cGY Day -1
  Stem cell infusion: Given Day 0
- Campath and TBI Conditioning (A2): Patients with sickle cell disease or thalassemia who do not have an HLA-identical sibling donor or who has pre-existing organ dysfunction making myeloablative condition ineligible will receive Campath on day -10 through -6, Cyclophosphamide on day -7, Fludarabine on day -6 through -2, total body irradiation (TBI) on day -1, stem cell infusion on Day 0.
  Campath, Fludarabine, Cyclophosphamide: Receives Campath-1H 0.2 mg/kg Days -10 through -6, Fludarabine 35 mg/m2 intravenous (IV) Days -6 through -2, total body irradiation (TBI) 300 cGy Day -1.
  Total Body Irradiation: 300 cGY Day -1
  Stem cell infusion: Given Day 0
Period: Overall Study
Arm/Group | Full Conditioning (Discontinued / A) | Busulfan Conditioning (B) | Campath and TBI Conditioning (A2)
Started | 3 | 5 | 14
Completed | 3 | 5 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Conditioning (Discontinued / A) | Busulfan Conditioning (B) | Campath and TBI Conditioning (A2) | Total
Number analyzed (Participants) | 3 | 5 | 14 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 5 | 12 | 20
  Between 18 and 65 years | 0 | 0 | 2 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 8 | 11
  Male | 1 | 4 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced Grade 3-5 Treatment Related Toxicity
Description: In general, grade 3 equates to moderate, grade 4 to severe and grade 5 to death.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 0 | 0 | 2

2. Secondary Outcome: The Incidence of Chimerism at 100 Days
Description: The number of patients whose blood and/or bone marrow contains > 10% donor cells.
Time Frame: 100 days
Population: One of the 3 patients treated on Arm A was retreated at Day 40 and was not evaluable. One of the 14 patients on Arm A2 died before 100 days.
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 2 | 5 | 13
Participants | 1 | 5 | 11

3. Secondary Outcome: The Incidence of Chimerism at 6 Months
Description: The number of patients whose blood and/or bone marrow contains > 10% donor cells.
Time Frame: 6 months
Population: One of the 3 patients treated on Arm A was retreated at Day 40 and was not evaluable. One of the 14 patients on Arm A2 died before 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 2 | 5 | 13
Participants | 1 | 5 | 8

4. Secondary Outcome: The Incidence of Chimerism at 1 Year
Description: The number of patients whose blood and/or bone marrow contains > 10% donor cells.
Time Frame: 1 year
Population: One of the 3 patients treated on Arm A was retreated at Day 40 and was not evaluable. One of the 14 patients on Arm A2 died before 1 year.
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 2 | 5 | 13
Participants | 1 | 5 | 8

5. Secondary Outcome: The Incidence of Grade 2-4 Acute Graft Versus Host Disease (Acute GVHD)
Description: The number of patients who experienced grades 2-4 Acute GVHD. Acute GVHD is when the donated bone marrow or peripheral blood stem cells view the recipient's body as foreign, and the donated cells/bone marrow attack the body. Grades 2-4 equate to mild to severe disease. Symptoms typically appear within weeks after transplant.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 0 | 0 | 0

6. Secondary Outcome: The Incidence of Grade 3-4 Acute Graft Versus Host Disease (Acute GVHD)
Description: The number of patients who experienced grades 3-4 Acute GVHD. Acute GVHD is when the donated bone marrow or peripheral blood stem cells view the recipient's body as foreign, and the donated cells/bone marrow attack the body. IGrades 3-4 equate to moderate to severe disease. Symptoms typically appear within weeks after transplant.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 0 | 0 | 0

7. Secondary Outcome: The Incidence of Chronic Graft Versus Host Disease (Chronic GVHD)
Description: The number of patients who experienced Chronic GVHD. Chronic GVHD is when the donated bone marrow or peripheral blood stem cells view the recipient's body as foreign, and the donated cells/bone marrow attack the body. Chronic GVHD can appear at any time after allogeneic transplant or several years after transplant.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 0 | 0 | 0

8. Secondary Outcome: The Incidence of Chronic Graft Versus Host Disease (Chronic GVHD)
Description: as for outcome 7
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 0 | 0 | 0

9. Secondary Outcome: Change in the Patient's Quality of Life as Compared to the Pre-Transplant Assessment
Description: The measure for quality of life used in this study is the Karnofsky Performance Score. The Karnofsky Performance Score runs from 100 to 0, where 100 is "perfect" health and 0 is death.
Time Frame: pre-transplant
Measure: Median (Full Range); unit: units on a scale
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
units on a scale | 100 [100 to 100] | 98 [90 to 100] | 99 [90 to 100]

10. Secondary Outcome: Change in the Patient's Quality of Life as Compared to the Pre-Transplant Assessment
Description: as for outcome 9
Time Frame: 1 year
Population: Two of the 14 patients treated on Arm A2 died before 1 year.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 12
units on a scale | 97 [90 to 100] | 100 [100 to 100] | 100 [80 to 100]

11. Secondary Outcome: Change in the Patient's Quality of Life as Compared to the Pre-Transplant Assessment
Description: as for outcome 9
Time Frame: 2 years
Population: Two of the 14 patients treated on Arm A2 died before 2 years and 2 failed their 2 year clinic appointment.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 10
units on a scale | 100 [90 to 100] | 100 [100 to 100] | 100 [90 to 100]

12. Secondary Outcome: Determine Physical Characteristics and Biologic Effects of Mixed Populations of Donor and Host Red Blood Cells
Time Frame: During study
Population: data were not collected
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Determine the Concentration of Campath in the Serum
Time Frame: Day 0
Population: The Principal Investigator removed this as a study objective and therefore Campath concentrations were not collected.
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Overall Survival
Description: Number of patients alive 100 days after transplant.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 3 | 5 | 12

15. Secondary Outcome: Overall Survival
Description: Number of patients alive 1 year after transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 3 | 5 | 12

16. Secondary Outcome: Disease Free Survival
Description: Number of patients alive without disease 100 days after transplant.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 3 | 5 | 11

17. Secondary Outcome: Disease Free Survival
Description: Number of patients alive without disease 1 year after transplant.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | RIC Bu/Flu (A) (Discontinued) | MA Bu/Cy (B) | RIC Cy/Flu/TBI (A2)
Number analyzed (Participants) | 3 | 5 | 14
Participants | 3 | 5 | 11

ADVERSE EVENTS:
Arm/Group | Full Conditioning (Discontinued / A) | Busulfan Conditioning (B) | Campath and TBI Conditioning (A2)
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/5 | 0/14
Other Adverse Events (participants affected / at risk) | 3/3 | 5/5 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Conditioning (Discontinued / A) (N=3) | Busulfan Conditioning (B) (N=5) | Campath and TBI Conditioning (A2) (N=14)
Primary Graft Failure (General disorders) | 1 | 0 | 0
Secondary Graft Failure (General disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Full Conditioning (Discontinued / A) (N=3) | Busulfan Conditioning (B) (N=5) | Campath and TBI Conditioning (A2) (N=14)
Bacterial Infection, Blood (Infections and infestations) | 2 | 2 | 5
Bacterial Infection, Pulmonary (Infections and infestations) | 0 | 1 | 2
Conjunctival Hemorrhage (Eye disorders) | 0 | 0 | 2
Delayed Growth/Stature (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Fungal Infection, Gastrointestinal (Infections and infestations) | 2 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 8
Hypothyroidism (Endocrine disorders) | 3 | 1 | 1
Pericardial Effusion (Cardiac disorders) | 0 | 3 | 3
Pneumonia (Infections and infestations) | 1 | 3 | 5
Renal Failure (Renal and urinary disorders) | 0 | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Second Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Seizure (Nervous system disorders) | 1 | 0 | 2
Veno-Occlusive Disease (Hepatobiliary disorders) | 0 | 0 | 2
Viral Infection, Blood (Infections and infestations) | 1 | 0 | 5
Viral Infection, Pulmonary (Infections and infestations) | 0 | 2 | 6
Cystitis (Renal and urinary disorders) | 1 | 1 | 1
Elevated Liver Function Tests (Investigations) | 1 | 0 | 0
Engraftment Syndrome (Immune system disorders) | 1 | 0 | 0
Esophageal Varices (Gastrointestinal disorders) | 0 | 0 | 1
Fungal Infection, Blood (Infections and infestations) | 1 | 0 | 1
Fungal Infection, Genitourinary (Infections and infestations) | 0 | 0 | 1
Fungal Infection, Pulmonary (Infections and infestations) | 0 | 0 | 1
Hemochromatosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hepatitis (Investigations) | 1 | 0 | 0
Hypogonadism (Endocrine disorders) | 1 | 0 | 1
Intraventricular Septal Hypertrophy (Cardiac disorders) | 0 | 0 | 1
Joint Dysfunction (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neuro Toxicity, NOS (Nervous system disorders) | 1 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 1 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 1
Paronychia of Bilateral Great Toes (Infections and infestations) | 0 | 0 | 1
Polycythemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Polymorphic Post-Transplant Lymphoproliferative Disorder (Blood and lymphatic system disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Subarachnoid Hemorrhage (Nervous system disorders) | 0 | 0 | 1
Thrombus, Right Atrium (Vascular disorders) | 0 | 0 | 1
Upper Respiratory Stridor (Reproductive system and breast disorders) | 1 | 0 | 0
Viral Infection, Gastrointestinal (Infections and infestations) | 0 | 2 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No